CLINICAL TRIAL: NCT07131423
Title: Effectiveness of Extracorporeal Shockwave Therapy Based on Fascial Manipulation Theory for Lateral Epicondylitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ZHANG PENG (Other)
Collaborators: Zhongda Hospital (Other)
Responsible Party: Sponsor-Investigator, ZHANG PENG, Chief Therapist, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025ZDSYLL214
Record Dates: First submitted 2025-08-11; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Lateral Epicondylitis (Tennis Elbow)
Keywords: Fascial Manipulation; Extracorporeal Shockwave Therapy; Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Active Comparator): Group A (Local ESWT): ESWT (2,500 impulses/session) at the lateral epicondyle point of maximal tenderness.
  Interventions: Device: Standard extracorporeal shock wave therapy
- Group B (Experimental): Group B (FM-guided ESWT): ESWT (2,500 impulses) at four Fascial Manipulation (FM)-selected Coordinating Centers (CCs) proximal to the epicondyle, with impulses weighted by tissue density.
  Interventions: Device: CC points shock wave therapy
- Group C (Experimental): Group C (Combined): Hybrid ESWT: 1,000 impulses at the epicondyle + 1,500 impulses at three FM-identified CCs.
  Interventions: Device: Shock wave therapy for the CC points and the lateral epicondyle

INTERVENTIONS:
Device: Standard extracorporeal shock wave therapy — ESWT was performed using the Swiss DolorClast Master ESWT device in accordance with the guidelines of the International Society of Medical Shockwave Therapy. The treatment was carried out by a physical therapist with at least 5 years of ESWT experience. The patient sat with the shoulder abducted at 45°, the elbow flexed at 90°, and the forearm supinated. The shock waves were delivered in a circular motion, targeting the 2-3 most painful tender points within a 3 cm radius centered on the lateral epicondyle. A total of 2,500 pulses were administered per session (0.2 to 2 bar, 8 Hz, 2,500 pulses, with intensity adjusted according to the patient's tolerance). All patients received a total of 4 ESWT sessions, once every 5 days, over a period of 3 weeks.
  Arms: Group A
Device: CC points shock wave therapy — The assessment was conducted by a 5-year or more experienced FM therapist, following the standard procedure of the FM organization. The process included conducting interviews, filling out assessment forms, performing movement checks, and conducting palpation. Four CC points covering the entire upper limb, including the shoulder area, were selected. The points were ranked based on the severity of the dense touch. The blackboard pen was used to mark the points on the patient's body. The same ESWT therapist as in Group A used the same shock wave treatment instrument to treat the four CC points. The most severe point received 800 shocks, the second most received 700 shocks, and the remaining two points each received 500 shocks. A total of 2,500 pulses (with an intensity of 0.2 to 2 bar, a frequency of 8 Hz, and the intensity adjusted according to the depth of the point and the patient's tolerance) were administered. This treatment was performed once every 5 days for 3 weeks.
  Arms: Group B
Device: Shock wave therapy for the CC points and the lateral epicondyle — Carry out the same process as Group B, but only select the three most severe CC points for shock therapy. Also, rank them according to the severity of the touch examination-induced densification. The most severe point receives 600 pulses, the second most severe receives 500 pulses, and the third most severe receives 400 pulses. At the same time, treat the lateral epicondylitis pain area in the same way as Group A. Apply 1000 pulses to the pain area. The total number of shocks for all treatments is 2500 (with an intensity of 0.2 to 2 bar, a frequency of 8 Hz, and the intensity is adjusted according to the depth of the point and the patient's tolerance). The therapist performing the treatment is the same as those in Group A and Group B. The treatment is carried out once every 5 days for 3 weeks.
  Arms: Group C

SUMMARY:
Goal:

This clinical trial aims to find out if using fascial theory to guide shockwave therapy works better for treating "tennis elbow" (pain on the outer side of the elbow) compared to standard shockwave treatment. It will also check for any side effects.

Main Questions:

Does treating fascial points (key tension areas in the arm) with shockwaves reduce pain more than just treating the elbow? Are there any temporary discomforts (like soreness or swelling) after treatment?

How It Works:

Researchers will compare three approaches:

Group A: Shockwaves applied only to the painful elbow area (standard treatment).

Group B: Shockwaves applied to 4 fascial points in the arm/shoulder (no elbow treatment).

Group C: Shockwaves applied to both the elbow and 3 fascial points.

Participants Will:

Receive 4 shockwave sessions (1 session every 5 days). Report pain levels, grip strength, and daily activities for 3 months. Attend follow-up visits to track progress.

Why It Matters:

If successful, this could lead to a more effective way to treat tennis elbow-by targeting the root cause of tension in the arm's connective tissue, not just the pain spot.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent pain at the lateral epicondyle of the humerus for ≥ 3 months
2. Pain is palpable at the lateral epicondyle of the humerus during examination
3. Positive Thompson's test (i.e., the patient reports pain when performing resisted extension while slightly extending the wrist joint, flexing the fist, extending the elbow joint, and having the forearm in an ulnar deviation position)
4. Positive Mill's test (i.e., the patient reports pain when performing resisted supination while slightly flexing the elbow joint, having the forearm in an ulnar deviation position, slightly extending the wrist joint, and flexing the fist)
5. Pain occurs during resisted extension of the index finger
6. Age between 18 and 65 years old. The participants in our study included those who were frequently active.

Exclusion Criteria:

* Tendon rupture, nerve root type cervical spondylosis, cubital or carpal tunnel syndrome, local infection, pregnancy, malignant tumor, bilateral tennis elbow, carpal tunnel syndrome, medial epicondylitis, elbow arthritis or instability, having systemic inflammatory diseases such as rheumatoid arthritis or ankylosing spondylitis, cognitive impairment making it difficult to cooperate, ipsilateral shoulder dysfunction, neurological abnormalities, radial nerve compression, arrhythmia or having a cardiac pacemaker implanted, diabetes, having received physical therapy and/or corticosteroid injections in the past three months.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Grip strength | Baseline, one week after all treatments, six weeks after all treatments, three months after all treatments.
  Participants will be required to adopt a shoulder-width stance, with their arms naturally hanging down and close to their bodies, and their elbows fully extended. The pain-free grip strength will be measured until pain occurs when the subject slowly squeezes the grip force gauge. The maximum grip strength will be measured at the maximum grip strength level. The average value of three consecutive trials will be calculated, with an interval of 20 seconds between each trial.
VAS(visual analogue scale) | Baseline, one week after all treatments, six weeks after all treatments, three months after all treatments.
  Pain intensity over the past week (at rest, during activity, and at night) was evaluated using a 0-10 cm horizontal visual analogue scale (VAS), where 0 represented no pain and 10 represented the most severe pain imaginable.
PRTEE(Patient-Rated Tennis Elbow Evaluation) | Baseline, one week after all treatments, six weeks after all treatments, three months after all treatments.
  Five items for pain (0 = no pain, 10 = the most severe pain imaginable) and physical function (six specific activity items and four daily activity items, 0 = no difficulty, 10 = unable to do), ranging from 0 to 100 points, with higher scores indicating more severe pain and greater functional loss.
PPT(pressure pain threshold) | Baseline, one week after all treatments, six weeks after all treatments, three months after all treatments.
  The PPT was evaluated at two sites, namely the lateral epicondyle of the humerus and 1 cm lateral to the lateral epicondyle. The patient was in a sitting position, with the shoulder externally rotated by 30°, the elbow flexed at 90°, and the forearm, wrist and hand supported on the table. Under this posture, the PPT measurement was conducted three times for each condition.

SECONDARY OUTCOMES:
Quick-DASH66 | Baseline, one week after all treatments, six weeks after all treatments, three months after all treatments.
  This questionnaire consists of eleven questions and uses a 5-point scale for scoring, similar to that of DASH. The total score and the scores of each module will be calculated on a 100-point scale, with higher scores indicating a worse condition. The reported minimum clinically important difference is 15.91 points.
Ultrasound shear wave elastography | Baseline, one week after all treatments, six weeks after all treatments, three months after all treatments.
  Each patient was required to sit in front of the examiner, with the elbows flexed at 90°, the thumb pointing upwards, and to maintain a relaxed forearm position throughout the measurement process. The transducer was placed vertically on the skin surface at the lateral epicondyle of the humerus, in contact with the skin surface slightly using a coupling agent to avoid compression effects. The CET attached to the lateral epicondyle of the humerus was scanned in the longitudinal plane (parallel to the direction of the CET fibers) to obtain standardized images.
Participant satisfaction | Baseline, one week after all treatments, six weeks after all treatments, three months after all treanments.
  The participants' satisfaction level with the progress of their condition will be determined using a validated 4-point Likert scale, ranging from "very satisfied", "somewhat satisfied", "somewhat dissatisfied" to "very dissatisfied".

CONTACTS AND LOCATIONS:
Overall Officials: MING MA, Study Director — Zhongda Hospital; Peng 张, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital Southeast University, Nanjin, Jiangsu, China